CLINICAL TRIAL: NCT02462382
Title: Efficacy of Continuous Infusion Ropivacaine Interscalene Blocks Versus Placebo for Pain Control After Arthroscopic Rotator Cuff Repair
Brief Title: Efficacy of Continuous Infusion Ropivacaine Interscalene Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Principal Investigator, Paula J. Harriott, Clinical Research Coordinator, Orlando Health, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13.121.08
Record Dates: First submitted 2015-05-28; First posted 2015-06-04 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: Full-thickness Rotator Cuff Tear
MeSH Terms: interventions — Ropivacaine; Drug Evaluation; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine infusion (Active Comparator): 270cc of Ropivacaine infusion at 5cc per hour. All patients will receive a reservoir for their catheters containing 280cc of either ropivacaine or saline that will infuse at a rate of 6cc per hour. The reservoirs will be attached in the operating room at the completion of the rotator cuff repair. Patients will be randomized intraoperative to receive either the ropivacaine or the saline.
  Interventions: Procedure: Arthroscopic Rotator Cuff Repair; Drug: Ropivacaine
- Saline infusion (Placebo Comparator): 270cc of Normal Saline infusion at 5cc per hour. All patients will receive a reservoir for their catheters containing 280cc of either ropivacaine or saline that will infuse at a rate of 6cc per hour. The reservoirs will be attached in the operating room at the completion of the rotator cuff repair. Patients will be randomized intraoperative to receive either the ropivacaine or the saline.
  Interventions: Procedure: Arthroscopic Rotator Cuff Repair; Drug: Saline

INTERVENTIONS:
Procedure: Arthroscopic Rotator Cuff Repair — During arthroscopic rotator cuff surgery, the surgeon inserts a small camera, called an arthroscope, into your shoulder joint. The camera displays pictures on a television screen, and your surgeon uses these images to guide miniature surgical instruments to repair the torn ligament.
  Other Names: Shoulder arthroscopy
Drug: Ropivacaine — The study group will receive a pump with study drug attached to a catheter placed into the shoulder area by the anesthesiologist.
  Other Names: Study drug
  Arms: Ropivacaine infusion
Drug: Saline — The control group will receive a pump with saine attached to a catheter placed into the shoulder area by the anesthesiologist.
  Other Names: Placebo
  Arms: Saline infusion

SUMMARY:
Arthroscopic rotator cuff repair is a common and painful procedure routinely performed on an outpatient basis. Postoperative pain control regimens can include narcotic pain medicine, non-steroidal anti-inflammatory medications and regional anesthesia such as an interscalene block (ISB). Regional blocks such as ISB can safely provide complete pain relief for the shoulder and upper extremity for eight to twelve hours1. However, the shoulder is still very painful when the block wears off. The purpose of this study is to:

1. Examine the efficacy of continuous infusion scalene block ropivacaine catheters during the first two days after arthroscopic rotator cuff repair.
2. Examine narcotic consumption after continuous infusion scalene block ropivacaine and placebo catheters after arthroscopic rotator cuff repair.
3. Evaluate for any continued pain relief benefit of continuous infusion scalene block ropivacaine catheters during the three days after the infusion catheters have finished.

DETAILED DESCRIPTION:
Patients undergoing arthroscopic rotator cuff repair by one of the three attending surgeon authors at Orlando Orthopaedic Outpatient Surgery Center will be candidates for the study. Further inclusion criteria will be a full-thickness rotator cuff tear, age eighteen or greater, a reparable rotator cuff tear and willingness to consent to study participation. Patients will not be excluded for concomitant procedures such as acromioplasty, distal clavicle resection, biceps tenotomy and biceps tenodesis.

Exclusion criteria will include age less than eighteen, irreparable rotator cuff tear, subscapularis tear requiring repair, labral tear requiring repair, allergy to ropivacaine or a similar local anesthetic agent and allergy to oxycodone.

All patients will undergo an ultrasound guided ISB with 30cc of 0.5% ropivacaine with epinephrine in the preoperative holding area by an anesthesiologist trained in regional block anesthesia. A continuous infusion catheter will be placed under ultrasound guidance to confirm appropriate position. An adhesive dressing on the skin will be used to keep the catheter in position and away from the operating field.

All patients will receive a reservoir for their catheters containing 280cc of either ropivacaine or saline that will infuse at a rate of 6cc per hour. The reservoirs will be attached in the operating room at the completion of the rotator cuff repair. Patients will be randomized intraoperative to receive either the ropivacaine or the saline. Randomization will be performed by block number randomization and the group assignments will be placed in sealed envelopes. The envelopes will be opened by the operating room circulating nurse. Both patients and surgeons will be blinded to the randomization.

Patients and their families will be educated preoperative and postoperative on the removal of the pain catheters. There will be written instructions regarding catheter removal. Patients or their family members will remove the catheters after the reservoirs are empty. The study authors will be available to assist with any catheter removal issues that the patients may have.

Patients will be prescribed oxycodone 5mg tablets for their postoperative pain control. Patients will receive diaries to record their pain levels utilizing visual analog scores (VAS) for the first five postoperative days. The first pain level will be recorded in the post anesthesia care unit. Pain levels will then be recorded twice daily. Patients will also be asked to log their oxycodone use during the first five postoperative days. Patients will be educated preoperative on the postoperative diaries. They will also receive a call from an OOOSC nurse on postoperative day one to address any questions or concerns.

Patients will be evaluated in the office by the operating surgeon at one week postoperative. At that time, study diaries will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for inclusion in the study if they have a full-thickness rotator cuff tear that has been deemed reparable by preoperative MRI. They will be included in the study if they are medically stable to undergo the surgery and consent to involvement in the study.

Exclusion Criteria:

1. Prior surgery on the involved shoulder
2. Preoperative MRI suggesting that the rotator cuff tear is irreparable
3. Patients with known allergies to oxycodone, ropivacaine or a similar drug
4. Workman's compensation patients
5. Patients who do not fill out their visual analog scores or their medication diaries
6. Patients with labral or subscapularis tears requiring repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2016-05-20 (Actual); Study Completion 2016-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randy Schwartzberg, MD, Principal Investigator — Orlando Orthopedic Center
Locations (1):
- Orlando Orthopaedic Center, Orlando, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects were asked to participate during their clinic visits.
Groups:
- Ropivacaine Infusion: 270cc of Ropivacaine infusion at 5cc per hour. All patients will receive a reservoir for their catheters containing 280cc of either ropivacaine or saline that will infuse at a rate of 6cc per hour. The reservoirs will be attached in the operating room at the completion of the rotator cuff repair. Patients will be randomized intraoperative to receive either the ropivacaine or the saline.
  Arthroscopic Rotator Cuff Repair: During arthroscopic rotator cuff surgery, the surgeon inserts a small camera, called an arthroscope, into your shoulder joint. The camera displays pictures on a television screen, and your surgeon uses these images to guide miniature surgical instruments to repair the torn ligament.
  Ropivacaine
- Saline Infusion: 270cc of Normal Saline infusion at 5cc per hour. All patients will receive a reservoir for their catheters containing 280cc of either ropivacaine or saline that will infuse at a rate of 6cc per hour. The reservoirs will be attached in the operating room at the completion of the rotator cuff repair. Patients will be randomized intraoperative to receive either the ropivacaine or the saline.
  Arthroscopic Rotator Cuff Repair: During arthroscopic rotator cuff surgery, the surgeon inserts a small camera, called an arthroscope, into your shoulder joint. The camera displays pictures on a television screen, and your surgeon uses these images to guide miniature surgical instruments to repair the torn ligament.
  Saline
Period: Overall Study
Arm/Group | Ropivacaine Infusion | Saline Infusion
Started | 24 | 27
Completed | 24 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine Infusion | Saline Infusion | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 26 | 49
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 15 | 18 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Mean Visual Analog Scale Score [Mean (Full Range); unit: Units on a scale] — Visual Analog Scale pain scale score 0-10. 0 equals no pain, 10 equals severe pain. Post Operation Day zero (POD 0) equals immediately after surgery. POD 1 equals the first day after surgery, POD 2 equals the second day after surgery. POD 3, all the way to POD 5 which is the 5th day after surgery.
  This study did not specifically compare patients based on incision/tear size. All attempts were made to locate the data but it is not available.
  Units on a scale
    POD 0 1cm incision | 0.3 [0 to 0.9] | 0 [0 to 0] | 0.3 [0 to 0.9]
    POD 0 2cm incision | 0.9 [0 to 1.7] | 0.8 [0.1 to 1.5] | 0.85 [0 to 1.5]
    POD 0 3cm incision | 0.23 [0 to 0.5] | 0.24 [0 to 0.5] | 0.23 [0 to 0.5]

OUTCOME MEASURES:

1. Primary Outcome: Mean Visual Analog Scale
Description: Shoulder Pain as measured by Visual Analog Scale, score 0-10. 0 equals no pain, 10 equals severe pain.
  Data not available for each tear size, all attempts were made to locate.
Time Frame: During the first two Post Operative Days.
Population: The study did not compare patients based on tear/incision size. All attempts were made to locate this data but it is unavailable.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ropivacaine Infusion | Saline Infusion
Number analyzed (Participants) | 24 | 27
units on a scale
  POD1 1cm incision | 3.5 [2.2 to 4.8] | 5.9 [5.0 to 6.9]
  POD 1 2cm incision | 3.1 [2.1 to 4.2] | 5.2 [4.3 to 6.1]
  POD 1 3cm incision | 4.0 [2.8 to 5.1] | 5.4 [4.4 to 6.3]
  POD 2 1cm incision | 2.9 [1.8 to 4.0] | 4.0 [3.0 to 4.9]
  POD 2 2cm incision | 3.1 [1.8 to 4.3] | 3.6 [2.5 to 4.7]
  POD 2 3 cm incision | 3.8 [2.8 to 4.9] | 4.1 [3.1 to 5.1]
Statistical Analysis 1: Comparison: Ropivacaine Infusion; Comparisons of pain scores using a Visual Analog Scale (VAS) based on Post-Operative Day (POD); Test type: Equivalence — The univariate analyses were conducted using Independent t-Tests for continuous variables and Fisher Exact Tests or Chi-Square Tests of Independence for categorical comparisons; p = .006, Chi-squared — POD 1 1cm incision; Fisher Exact Tests = .041

2. Secondary Outcome: Mean Visual Analog Scale Score
Description: Visual Analog Scale pain scale score 0-10. 0 equals no pain, 10 equals severe pain.
Time Frame: Post Operative Days (POD) 3, 4 and 5.
Population: All attempts were made to locate the data for the number of participants with different incision/tear sizes, but the data are not available.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ropivacaine Infusion | Saline Infusion
Number analyzed (Participants) | 24 | 27
units on a scale
  POD 3 1cm incision | 3.5 [2.3 to 4.6] | 3.3 [2.3 to 4.3]
  POD 3 2cm incision | 3.3 [2.2 to 4.4] | 3.1 [2.4 to 4.4]
  POD 3 3cm incision | 3.2 [2.2 to 4.2] | 3.4 [2.4 to 4.4]
  POD 4 1 cm incision | 2.6 [1.6 to 3.7] | 3.5 [2.5 to 4.5]
  POD 4 2cm incision | 2.6 [1.5 to 3.7] | 3.2 [2.3 to 4.1]
  POD 4 3cm incision | 2.8 [1.6 to 4.1] | 3.3 [2.4 to 4.3]
  POD 5 1cm incision | 2.3 [1.4 to 3.2] | 3.0 [2.1 to 3.9]
  POD 5 2cm incision | 2.2 [1.2 to 3.2] | 2.6 [1.7 to 3.5]
  POD 5 3cm incision | 2.8 [1.7 to 3.8] | 3.0 [2.0 to 4.0]

3. Secondary Outcome: Oxycodone Consumption
Time Frame: Post operative days 1 and 2.
Measure: Mean (Full Range); unit: Pills
Arm/Group | Ropivacaine Infusion | Saline Infusion
Number analyzed (Participants) | 24 | 27
Pills
  POD 1 | 5.8 [4.1 to 7.5] | 8.3 [6.6 to 10.0]
  POD 2 | 5.8 [4.1 to 7.6] | 7.9 [6.2 to 9.5]

4. Secondary Outcome: Oxycodone Consumption After the First Two Postoperative Days.
Time Frame: Post Operative Days 3, 4 and 5.
Measure: Mean (Full Range); unit: Pills
Arm/Group | Ropivacaine Infusion | Saline Infusion
Number analyzed (Participants) | 24 | 27
Pills
  POD 3 | 5.5 [3.9 to 7.0] | 5.8 [4.2 to 7.5]
  POD 4 | 3.9 [2.6 to 5.1] | 4.7 [3.2 to 6.2]
  POD 5 | 3.6 [2.4 to 4.8] | 3.7 [2.4 to 5.1]

ADVERSE EVENTS:
Time Frame: Each patient will be part of the study for a period of five days postoperatively. Adverse event data will be collected from the time of consent until 5 days post op.
Arm/Group | Ropivacaine Infusion | Saline Infusion
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 0/24 | 0/27

LIMITATIONS AND CAVEATS:
This study did not specifically compare patients based on incision size/tear size. Pain scores were never compared between tear size or incision size groups. All attempts were made to locate the data but it is not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No